CLINICAL TRIAL: NCT05940402
Title: A Phase 1 Open-label Trial to Evaluate the Pharmacokinetics and Safety Following a Single Dose of Emraclidine in Adult Participants With Mild, Moderate, and Severe Renal Impairment Compared With Adult Participants With Normal Renal Function
Brief Title: A Study to Evaluate Pharmacokinetic and Safety Trial of Emraclidine in Participants With Renal Impairment Compared With Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-SP-1007
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild Renal Impairment (Experimental): Participants will receive a single oral dose of 10 milligrams (mg) emraclidine on Day 1.
  Interventions: Drug: Emraclidine
- Moderate Renal Impairment (Experimental): Participants will receive a single oral dose of 10 mg emraclidine on Day 1.
  Interventions: Drug: Emraclidine
- Severe Renal Impairment (Experimental): Participants will receive a single oral dose of 10 mg emraclidine on Day 1.
  Interventions: Drug: Emraclidine
- Normal Renal Function (Experimental): Participants will receive a single oral dose of 10 mg emraclidine on Day 1.
  Interventions: Drug: Emraclidine

INTERVENTIONS:
Drug: Emraclidine — Oral tablets
  Other Names: CVL-231

SUMMARY:
The primary purpose of this study is to assess the effect of renal impairment on the pharmacokinetics (PK) of emraclidine following administration of a single oral dose in participants with mild, moderate, and severe renal impairment relative to matched participants with normal renal function.

ELIGIBILITY:
Key Inclusion Criteria:

1. For All Participants

   * Body mass index of ≥18.0 to 42.0 kilograms per meter square (kg/m^2), inclusive, and a total body weight ≥50 kilograms (kg) (110 pounds [lbs]).
   * Sexually active women of childbearing potential must agree to use at least an acceptable birth control method during the trial and for 7 days after the last dose of investigational medicinal product (IMP).
2. Additional Criteria for Participants With Normal Renal Function

   * Age that is within ±10 years of the median age for the renal impairment groups.
   * Body weight that is within ±15% of the median body weight for the renal impairment groups.
   * Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
   * Normal renal function: Estimated glomerular filtration rate (eGFR) ≥90 milliliter per minute (mL/min) determined using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. Renal function assessed at Baseline (Check-in/Day -1) should not deviate more than 30% from the Screening value.
3. Additional Criteria for Participants With Renal Impairment

   * Mild, moderate, or severe renal impairment based on eGFR determined using the 2021 CKD-EPI equation. Renal function assessed at Baseline (Check-in/Day -1) should not deviate more than 30% from the Screening value.
   * Stable disease, defined as no clinically significant changes in disease status as documented by most recent eGFR assessment (within at least 3 months before Screening).
   * Stable concomitant medications for the management of individual participant's medical history; on a case-by-case basis, with input from the sponsor, participants receiving fluctuating concomitant medication/treatment may be considered if the underlying disease is under control.

Key Exclusion Criteria:

1. For All Participants

   * "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

     * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
     * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
     * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
     * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
     * Suicidal Ideation Item 1 (Wish to be Dead)
     * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Any "yes" response on Suicidal Ideation Item 1 or Item 2 that was within the individual's lifetime but not within the past 12 months should be discussed with the medical monitor prior to inclusion of the participant in the trial.
   * Serious risk of suicide in the opinion of the investigator is also exclusionary.
   * History of moderate to severe substance or alcohol-use disorder (excluding nicotine or caffeine) as per DSM-5 criteria within 12 months prior to signing the informed consent form (ICF).
   * Receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination or booster within 7 days of planned dosing.

   In addition, participants who plan to receive SARS-CoV-2 vaccination or booster while participating in the trial or for a minimum of 7 days (to cover at least 5 half-lives of IMP) after the last dose of investigational medicinal product (IMP) will be excluded.

   - Have recently been diagnosed with symptomatic coronavirus disease-2019 (COVID-19) or test positive (i.e., using polymerase chain reaction [PCR] or rapid antigen test) for SARS-CoV-2 within 15 days prior to signing the ICF.
2. Additional Criteria for Participants With Normal Renal Function

   - Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for surgically excised non-melanomatous skin cancers or in situ cervical cancer, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
3. Additional Criteria for Participants With Renal Impairment

   * Evidence of disease that is not explained by current/known medical history, i.e., organ dysfunction (including malignancies) or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with renal impairment and other underlying conditions.
   * Participants who have received an organ transplant or are currently waiting for an organ transplant and are listed on the national transplant list.
   * Participants who require dialysis
   * Participants with nephrotic syndrome.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5
Maximum Observed Unbound Plasma Concentration (Cmax,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5
Area Under the Plasma Concentration-time Curve from Time Zero to t (AUC0-t) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5
Area Under the Unbound Plasma Concentration-time Curve from Time Zero to t (AUC0-t,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5
Area Under the Unbound Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 5

SECONDARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Up to Day 15
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 5
Number of Participants With Clinically Significant Changes in Vital Signs | Up to Day 5
Number of Participants With Clinically Significant Change in Laboratory Assessments | Up to Day 5
Number of Participants With Clinically Significant Change in Physical and Neurological Examination Results | Up to Day 5
Changes in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Day 5
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Tustin, California, Tustin, California
  - Miami, Florida, Miami, Florida
  - Orlando, Florida, Orlando, Florida
  - Knoxville, Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No